CLINICAL TRIAL: NCT01240876
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending-Dose Study to Evaluate the Safety and Efficacy of CEP-37247 Administered at Single Doses of 0.5, 1, 3, 6, or 12 mg by the Transforaminal Epidural Route for the Treatment of Patients With Lumbosacral Radicular Pain Associated With Disk Herniation
Brief Title: Study to Evaluate the Safety and Efficacy of Placulumab (CEP-37247) Administered by the Transforaminal Epidural Route for the Treatment of Patients With Lumbosacral Radicular Pain Associated With Disk Herniation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C37247/1083
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Sciatica
Keywords: Sciatica; Pain
MeSH Terms: conditions — Sciatica; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- CEP-37247 (Experimental)
  Interventions: Drug: CEP-37247
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CEP-37247 — 0.5-, 1-, 3-, 6-, and 12-mg doses of CEP-37247 will be administered by the transforaminal epidural route.
  Other Names: placulumab
  Arms: CEP-37247
Drug: Placebo — Matching placebo vials will be filled with the buffered solution for CEP-37247.
  Arms: Matching placebo

SUMMARY:
The primary objective of the study is to evaluate the safety and efficacy of CEP-37247 compared with placebo as assessed by the occurrence of adverse events, and the mean change in average pain intensity (API) in the affected leg.

ELIGIBILITY:
Inclusion Criteria:

* Over the 4 days prior to the randomization visit, the patient has a mean score greater than or equal to 5 (of 10) for "Average Pain Over the Past 24 Hours" for the pain in the affected leg as assessed by the 11-Point Numerical Rating Scale (NRS-11) captured in the electronic diaries. The patient must have valid (non-missing) data for at least 3 out of the 4 days, and the mean score must be at least 5 without rounding.
* The patient has a current diagnosis of lumbosacral radicular pain. Pain must radiate into the leg in a dermatomal/myotomal distribution consistent with the diagnosis of lumbosacral radicular pain in the suspected involved nerve root. Based on history and medical records (if available), the duration of the current episode of pain must be between 6 and 52 weeks duration.
* Diagnosis must be confirmed by magnetic resonance imaging (MRI) (or existing computed tomography [CT] or MRI related to the symptoms present at screening) performed within 6 months prior to screening and demonstrating disk herniation at a location consistent with the clinical symptoms of radicular pain. Other incidental pathology is permitted as long as it is asymptomatic and believed not causal of the primary diagnosis of lumbosacral radicular pain at the specific spinal level as described below.
* The patient must have at least 1 of the following: a positive straight leg raise (L5-S1), positive femoral stretch test (L3-L4), or other positive test result upon physical examination that is consistent with the presence of nerve root irritation at the nerve root suspected to be involved in the diagnosed lumbosacral radicular pain at screening.
* Herniation must affect L3-L4, L4-L5, or L5-S1 and must be consistent with clinical presentation of the current episode of lumbosacral radicular pain as described above.
* Patients with significant or progressive sensory impairment or motor impairment (such as foot drop) must be assessed on a case-by-case basis by the investigator, and must in each case receive written approval of the Sponsor prior to randomization.
* There must be confirmation that the patient does not have an active tuberculosis infection at screening. The patient should have either a negative QuantiFERON®-TB Gold blood test or negative tuberculin skin test (TST) result at screening; however if QuantiFERON®-TB Gold test or TST is positive, a chest radiogram may be used to determine whether a patient has an active infection.
* The patient is willing to keep all analgesic medication and other therapy usage (such as physiotherapy, acupuncture, or transcutaneous electrical nerve stimulation [TENS]) stable or decreased during the study and use only the rescue pain medication as needed and as specified by the protocol.
* The patient is in good health (with the exception of the condition under study) as determined by a medical and psychiatric history, medical examination, ECG, serum chemistry, hematology, urinalysis, and serology.
* Women of childbearing potential (ie, not surgically sterile or 2 years postmenopausal), must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study, and have a negative pregnancy test at screening.

Exclusion Criteria:

The patient:

* has a documented history of an allergic reaction (hives, rash, etc.) or a clinically significant intolerance to study drug or ingredients.
* has a body mass index (BMI) greater than 40 kg/m2.
* the patient has an established history of a major psychiatric disorder, not controlled with medication or appears to have anxiety that would interfere with clinical pain scores or participation in the trial.
* has clinically significant abnormalities in clinical chemistry, hematology or urinalysis, including serum glutamic-oxaloacetic transaminase/aspartate aminotransferase (AST) or serum glutamic-pyruvic transaminase/alanine aminotransferase (ALT) greater than or equal to 3 times the upper limit of the reference range or an estimated glomerular filtration rate (eGFR) less than or equal to 30 mL/min/1.73 m2 (Modification of Diet in Renal Disease [MDRD] study formula) at screening.
* has received an intra-epidural steroid injection for the treatment of the current episode of sciatica during the last 3 months prior to screening.
* has significant pain unrelated to the disk herniation that would significantly compromise assessment of the radicular back and leg pain related to the disk herniation.
* has radiologic evidence of disk herniation at more than 1 spinal level, and clinical evidence of lumbosacral radicular pain at more than 1 spinal nerve corresponding to the levels of the multiple disk herniations.
* has received any investigational drug within 30 days prior to screening, or is scheduled to receive an investigational drug other than blinded study drug during the course of this study.
* has had lumbar or sacral back surgery related to the specific disk that is the cause of the radicular pain upon presentation to the study, or currently plans to undergo spine surgical intervention while in the study.
* has received epidural corticosteroid injections in the back within 3 months of screening.
* is involved in an ongoing worker's compensation claim, disability claim, or litigation related to any pain problem.
* has any active infection that is not self-limiting and not resolved prior to study drug administration.
* has a history of malignancy or evidence of malignancy or lymphoproliferative or neoplastic disease with the exception of successfully treated basal or squamous cell carcinoma of the skin or cervical intraepithelial neoplasia within 5 years of the screening visit.
* has a history of systemic fungal infection.
* has a history of opportunistic infection within 3 months prior to screening.
* has a history of known or suspected chronic infection, tuberculosis, hepatitis B virus (HBV), hepatitis C virus (HCV), or Human Immunodeficiency Virus (HIV). The investigator will review all medical history (including medication history), and patients found to be HIV positive based on medical review are to be excluded from the study.
* has a history of any demyelinating disease, including multiple sclerosis and optic neuritis.
* has used anti-tumor necrosis factor (TNF) receptor medication (anakinra [KINERET®, Biovitrum]) or anti-TNF medication (etanercept [ENBREL®, Amgen Inc.], infliximab [REMICADE®, Centocor Ortho Biotech Inc.], or adalimumab [HUMIRA®, Abbott Laboratories], or any experimental TNF inhibitor) within the past year.
* has a planned joint replacement surgery or a history of infected joint prosthesis or has received antibiotics for a suspected infection of a joint prosthesis if that prosthesis has not been removed or replaced.
* has been given live vaccines within 14 days of study drug administration.
* has severe spinal stenosis or spondylolisthesis (grade 2 or higher).
* has coagulopathy.
* is a pregnant or lactating woman (any women becoming pregnant during the study will be withdrawn from the study).
* has a history of diabetic neuropathy or peripheral neuropathy in the lower extremities.
* has a history of any condition (not otherwise specified) known to be amenable to TNF inhibitors (e.g., Crohn's disease).
* has a known allergy or idiosyncratic (atopic) reaction to contrast agent, local anesthetic, study drug, any ingredient listed as being present in a study formulation, or any other pain management compound likely to be prescribed in the study, including their metabolites (if applicable) or any ingredient listed as being present in their formulations.
* has any clinically significant uncontrolled medical condition (treated or untreated).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events compared to placebo | throughout the 28-week double-blind treatment period
Mean change in the weekly average of daily average pain intensity (API) in the affected leg on the 11-Point Numerical Rating Scale (NRS-11) | at week 4 compared with baseline
  The average pain intensity over the past 24 hours on the NRS-11 will be collected daily by electronic diary.

SECONDARY OUTCOMES:
Weekly average of daily leg API score as assessed by the NRS-11 from electronic diary entries | at each of the first 6 weeks
  Evaluate the efficacy of each dose of CEP-37247 as compared with placebo within each individual dose group and with the combined placebo group.
Weekly average of daily back API score as assessed by the NRS-11 from electronic diary entries | at each of the first 6 weeks
  Evaluate the efficacy of each dose of CEP-37247 as compared with placebo within each individual dose group and with the combined placebo group.
Weekly average of daily worst leg pain score as assessed by the NRS-11 from electronic diary entries | at each of the first 6 weeks
  Evaluate the efficacy of each dose of CEP-37247 as compared with placebo within each individual dose group and with the combined placebo group.
Weekly average of daily worst back pain score as assessed by the NRS-11 from electronic diary entries | at each of the first 6 weeks
  Evaluate the efficacy of each dose of CEP-37247 as compared with placebo within each individual dose group and with the combined placebo group.
Patients with 30% and 50% reductions in average pain over the previous 24 hours as measured by the Brief Pain Inventory Short Form (BPI-SF) | at 1, 2, 4, 6, 14, and 28 weeks
  Evaluate the efficacy of each dose of CEP-37247 as compared with placebo within each individual dose group and with the combined placebo group.
Change in total Oswestry Disability Index (ODI) score as well as subscale scores | at 1, 2, 4, 6, 14, and 28 weeks
  Evaluate the efficacy of each dose of CEP-37247 as compared with placebo within each individual dose group and with the combined placebo group.
Score on the Patient Global Impression of Change | at 1, 2, 4, 6, 14, and 28 weeks
  Evaluate the efficacy of each dose of CEP-37247 as compared with placebo within each individual dose group and with the combined placebo group.
Change in 36-Item Short Form Health Survey (SF-36) score | from baseline to weeks 4, 14, and 28
  Evaluate the efficacy of each dose of CEP-37247 as compared with placebo within each individual dose group and with the combined placebo group.
Average daily amount of rescue medication used | during each of the first 6 weeks of the 28-week double-blind treatment period
  Evaluate the efficacy of each dose of CEP-37247 as compared with placebo within each individual dose group and with the combined placebo group.
Patients requiring a subsequent injection of epidural steroids | up to 28 weeks after CEP-37247 treatment
  Evaluate the efficacy of each dose of CEP-37247 as compared with placebo within each individual dose group and with the combined placebo group.
Patients requiring back surgery | up to 28 weeks after CEP-37247 treatment
  Evaluate the efficacy of each dose of CEP-37247 as compared with placebo within each individual dose group and with the combined placebo group.
Evaluate the safety of CEP-37247 treatment as assessed by vital signs measurements | at weeks 1, 2, 4, 6, 14, and 28 (or early termination)
Evaluate the safety of CEP-37247 treatment as assessed by electrocardiogram (ECG) results | at week 4
Evaluate the safety of CEP-37247 treatment as assessed by clinical laboratory tests | at weeks 1, 2, 4, 6, 14, and 28 (or early termination)
Evaluate the safety of CEP-37247 treatment as assessed by physical examination | at weeks 4 and 28 (or early termination)
Evaluate the safety of CEP-37247 treatment as assessed by neurologic examination | at weeks 1, 2, 4 and 28 (or early termination)
Evaluate the safety of CEP-37247 treatment as assessed by concomitant medication usage | throughout the 28-week double-blind treatment period
Evaluate the safety of CEP-37247 treatment as assessed by immunogenicity tests | at weeks 2, 4, 6, 14, and 28 (or early termination)
Characterize the serum pharmacokinetics of CEP-37247 following epidural administration | Throughout the 28-week double-blind treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Associate Director, Clinical Research, MD, PhD, Study Director — Cephalon
Locations (24):
- United States (20):
  - Teva Investigational Site 22, La Mesa, California
  - Teva Investigational Site 18, Laguna Hills, California
  - Teva Investigational Site 19, Pasadena, California
  - Teva Investigational Site 2, Pasadena, California
  - Teva Investigational Site 14, Orlando, Florida
  - Teva Investigational Site 5, Sarasota, Florida
  - Teva Investigational Site 10, Marietta, Georgia
  - Teva Investigational Site 13, Marietta, Georgia
  - Teva Investigational Site 9, Bloomington, Illinois
  - Teva Investigational Site 15, Overland Park, Kansas
  - Teva Investigational Site 8, Shreveport, Louisiana
  - Teva Investigational Site 20, Winston-Salem, North Carolina
  - Teva Investigational Site 16, Dayton, Ohio
  - Teva Investigational Site 21, Eugene, Oregon
  - Teva Investigational Site 17, Altoona, Pennsylvania
  - Teva Investigational Site 1, Greenville, South Carolina
  - Teva Investigational Site 11, North Charleston, South Carolina
  - Teva Investigational Site 6, Spartanburg, South Carolina
  - Teva Investigational Site 4, Orem, Utah
  - Teva Investigational Site 3, Salt Lake City, Utah
- Australia (4):
  - Teva Investigational Site 103, Caulfied South
  - Teva Investigational Site 102, Malvern East
  - Teva Investigational Site 100, North Terrace
  - Teva Investigational Site 101, St Leonards